CLINICAL TRIAL: NCT02641002
Title: A Phase 1, Open-label, Dose Finding Study of CC-90002, a Monoclonal Antibody Directed Against CD47, in Subjects With Acute Myeloid Leukemia and High-Risk Myelodsplastic Syndrome
Brief Title: A Study of CC-90002 in Subjects With Acute Myeloid Leukemia (AML) and High-risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preliminary monotherapy data in relapsed/refractory AML and high-risk MDS did not offer a sufficiently encouraging profile for further dose escalation/expansion
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90002-AML-001
Record Dates: First submitted 2015-11-12; First posted 2015-12-29 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: CC-90002; Monoclonal; Antibody; CD47; Hematologic Cancers; Acute Myeloid Leukemia; AML; Myelodysplastic syndrome; MDS; Blood disorder
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Diseases | interventions — CC-90002

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation of CC-90002 (Experimental): CC-90002 by intravenous (IV) infusion on a 28 day cycle
  Interventions: Drug: CC-90002

INTERVENTIONS:
Drug: CC-90002 — Monoclonal Ab to CD47

SUMMARY:
Study CC-90002-AML-001 is an open-label, Phase 1 dose escalation (Part A) and expansion (Part B), clinical study of CC-90002, administered by intravenous (IV) infusion, in subjects with relapsed and/or primary refractory AML and high-risk MDS. The study will explore escalating doses of CC-90002 using a 3 + 3 dose escalation design in Part A, followed by dose expansion in Part B.

The primary objective is to determine the safety and tolerability of CC-90002 and also to define the non-tolerated dose (NTD), the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of CC-90002.

DETAILED DESCRIPTION:
In both Part A and Part B, treatments will be administered in two phases starting with an induction phase followed by a maintenance phase. During the induction phase, treatments will be administered in 42-day cycles in Cycles 1 through 4. Following completion of Cycle 4 in the induction phase, subjects with non-progressive disease will enter the maintenance phase. During the maintenance phase, treatments will be administered in 28 day cycles. Subjects may continue CC-90002 for up to a maximum of 2 years (eg, induction phase Cycles 1 through 4 and maintenance phase Cycles 5 through 24) or until clinically significant disease progression, the occurrence of intolerable toxicity, or physician/subject decision to discontinue CC-90002, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age, at the time of signing the informed consent form (ICF).
2. Relapsed and/or primary refractory Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) with subtype refractory anemia with excess blasts (RAEB)-2 defined as high or very high-risk that is recurrent or refractory, or the patient is intolerant to established therapy.
3. Subject consents to hospitalization for first (Cycle 1 Day 1) dose of CC-90002 and for 72 hours after.
4. Subject consents to serial bone marrow aspiration and biopsies as specified.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2.
6. Eligible study subjects must exhibit acceptable liver, renal, and coagulation function as assessed by laboratory tests.
7. Females and males must practice true abstinence or agree to contraceptive methods throughout the study, and for up to 8 weeks following the last dose of CC 90002.

Exclusion Criteria:

1. Active central nervous system (CNS) leukemia or known CNS leukemia.
2. Immediately life-threatening, severe complications of leukemia.
3. Impaired cardiac function or clinically significant cardiac diseases.
4. Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
5. Prior autologous hematopoietic stem cell transplant ≤ 3 months.
6. Prior allogeneic hematopoietic stem cell transplant (HSCT) with either standard or reduced intensity conditioning ≤ 6 months.
7. Systemic immunosuppressive therapy post HSCT or with clinically significant graft-versus-host disease (GVHD).
8. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks whichever is shorter.
9. Major surgery ≤ 2 weeks and recovered from any clinically significant effects of recent surgery.
10. Pregnant or nursing females.
11. Known HIV infection.
12. Known chronic hepatitis B or C (HBV/HCV) infection.
13. Ongoing treatment with chronic, therapeutic dosing of anti-coagulants.
14. History of autoimmune hemolytic anemia or autoimmune thrombocytopenia.
15. History of concurrent second cancers requiring active, ongoing systemic treatment.
16. Subjects for whom potentially curative anticancer therapy is available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | Up to 26 months
  Number of participants with a DLT
Non-tolerated Dose (NTD) | Up to 26 months
  The NTD is defined as the dose at which 2 or more of up to 6 evaluable subjects in a cohort experience a DLT in Cycle 1
Maximum tolerated dose (MTD) | Up to 26 months
  The MTD is defined as the last dose level(s) below the NTD with 0 or 1 out of 6 evaluable subjects experiencing a DLT during Cycle 1.

SECONDARY OUTCOMES:
Preliminary Efficacy of CC-90002 | Up to 35 months
  Determined by response rates of acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) by disease-appropriate response criteria.
Pharmacokinetics-Cmax | Up to 35 months
  Maximum observed concentration in serum
Pharmacokinetics-AUC | Up to 35 months
  Area under the serum concentration - time curve
Pharmacokinetics-Tmax | Up to 35 months
  Time to peak (maximum) serum concentration
Pharmacokinetics-T 1/2 | Up to 35 months
  Terminal half-life (T 1/2)
Pharmacokinetics- CL | Up to 35 months
  Total body clearance of the drug from the serum
Pharmacokinetics- Vss | Up to 35 months
  Volume of distribution at steady-state
Anti-Drug Antibodies (ADAs) | Up to 35 months
  Determine the presence and frequency of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burgess, MD, PhD, Study Director — Celgene Corporation
Locations (6):
- United States (6):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - UCLA Division of Hematology Oncology, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Narla RK, Modi H, Bauer D, Abbasian M, Leisten J, Piccotti JR, Kopytek S, Eckelman BP, Deveraux Q, Timmer J, Zhu D, Wong L, Escoubet L, Raymon HK, Hariharan K. Modulation of CD47-SIRPalpha innate immune checkpoint axis with Fc-function detuned anti-CD47 therapeutic antibody. Cancer Immunol Immunother. 2022 Feb;71(2):473-489. doi: 10.1007/s00262-021-03010-6. Epub 2021 Jul 10. PMID 34247273